CLINICAL TRIAL: NCT05359497
Title: Value of MRCP+ And Liver Multiscan in the Management of Dominant Strictures in Primary Sclerosing Cholangitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Perspectum (Industry)
Responsible Party: Principal Investigator, C.Y. Ponsioen, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MALD study
Record Dates: First submitted 2022-03-23; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: PSC; MRI
Keywords: Liver Multiscan; MRCP+
MeSH Terms: interventions — Cholangiopancreatography, Magnetic Resonance

STUDY DESIGN:
Intervention Model Description: Prospective, observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Additional sequences and extra MRI (Other): PSC patients, suspected for having a dominant stenosis, that undergo additional LMS sequences next to standard care MRI prior to ERCP and an additional MRI/MRCP with additional LMS sequences 8 weeks after ERCP.
  MRI images will be analysed by the post-processing tool called MRCP+ and Liver Multiscan, which are performed after the MRI is performed.
  Interventions: Diagnostic Test: Liver Multiscan sequences baseline; Device: MRCP+ analysis baseline; Device: Liver Multiscan analysis baseline; Diagnostic Test: MRI liver with MRCP; Diagnostic Test: Liver Multiscan sequences follow-up; Device: MRCP+ analysis follow up; Device: Liver Multiscan analysis follow up

INTERVENTIONS:
Diagnostic Test: Liver Multiscan sequences baseline — Additional Liver Multiscan sequences at baseline besides standard care MRI liver /MRCP prior to ERCP.
Device: MRCP+ analysis baseline — Post processing tool (Software) for quantifying MRCP images after MRCP is performed. Patient involvement is not necessary during this procedure.
Device: Liver Multiscan analysis baseline — Post processing tool (Software) for determining the corrected T1 time after the additional LMS sequences at baseline are performed. This cT1 reflects the activity of inflammation/fibrosis of the liver. Patient involvement is not necessary during this procedure.
  Other Names: LMS
Diagnostic Test: MRI liver with MRCP — An extra MRI liver with contrast and MRCP is performed 8 weeks after the ERCP following standard care protocol
Diagnostic Test: Liver Multiscan sequences follow-up — Additional Liver Multiscan sequences are performed at 8 weeks after ERCP.
Device: MRCP+ analysis follow up — Post processing tool (Software) for quantifying MRCP images after the MRCP from follow up is performed. Patient involvement is not necessary during this procedure.
Device: Liver Multiscan analysis follow up — Post processing tool (Software) for determining the corrected T1 time after the additional LMS sequences from the follow up scan are performed. This cT1 reflects the activity of inflammation/fibrosis of the liver. Patient involvement is not necessary during this procedure.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a chronic progressive biliary disease. Due to the heterogeneous disease course and the relatively low clinical event rate of 5% per year it is difficult to predict prognosis of individual patients. Novel imaging techniques called MRCP+ and Liver Multiscan (LMS) hold the prospect of adequate depicting and quantifying lesions of the biliary tree as well as capturing functional derailment. However, these features must be tested first.

The purpose of this study is to assess the (i) ability of MRCP+ to detect change in biliary volume, (ii) reproducibility of MRCP+ and LMS, and (iii) correlation of MRCP+ with ERC findings as gold standard.

DETAILED DESCRIPTION:
After informed consent, patients will undergo standard care with blood tests and MRI/MRCP. While performing the MRI, additional sequences called LMS are performed. Thereafter, an ERCP will be performed. Approximately 8 weeks after ERCP, another MRI/MRCP and LMS will be performed. Also, blood tests will be performed and a clinician will evaluate the clinical condition and complaints of patients

Images will be coded and analysed by Perspectum to retrieve MRCP+ and LMS results.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis according to the IPSCSG Definitions (22)
* Age ≥ 18
* Able to give informed consent
* Clinically suspicious for a dominant stricture

Exclusion Criteria:

* insufficient image quality
* known allergy for MRI contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in total biliary volume by MRCP+ and cT1 by LMS 8 weeks after endoscopic treatment of dominant strictures | 1st MRI: Baseline = week 0. 2nd MRI: week 8 after ERCP
  Decrease in total biliary volume (in ml, measured by MRCP+) and decrease in cT1 (in ms, measured by LiverMultiscan), which will be assessed by performing paired t-tests.

SECONDARY OUTCOMES:
Correlation of MRCP+/Liver Multiscan with the modified Amsterdam cholangiographic classification | 1st MRI: Baseline = week 0. 2nd MRI: week 8 after ERCP
  The outcomes of both MRCP+ and Liver Multiscan of the baseline MRI will be compared with the modified amsterdam cholangiographic classification and the correlation coefficient will be calculated. The cholangiographic classification uses age and classification of the intrahepatic and extrahepatic biliary ducts to determine a prognostic score. This score ranges from 0-40, in which a score of 40 reflects the worst prognosis with e.g. a 1-year survival of 29% and 5-year survival of 3.3%, while zero points reflect a 1-year or 5-year survival of 98% or 94%, respectively.
Correlation of imaging features of MRCP+ with classic cholangiography in individual areas of interest by two independent assessors. | 1st MRI: Baseline = week 0. 2nd MRI: week 8 after ERCP
  MRCP+ given dilatations and strictures are compared with the in-depth assessment of strictures and dilatations of the MRCP, by two independent radiologists, specialized in MRCP. The correlation coefficient will be calculated.
Correlation of dominant strictures rated by MRCP+/Liver Multiscan with those assessed by classic definition of dominant strictures. | 1st MRI: Baseline = week 0. 2nd MRI: week 8 after ERCP
  MRCP+ given strictures with increased liver multiscan values are compared with the assessment (by the hand of the classic definition) of strictures found on MRCP images. The assessment is performed by two independent radiologists, specialized in MRCP. The correlation coefficient will be calculated.
Repeated detection of dominant strictures, as determined by two independent assessors, that were not treated by ERC | 1st MRI: Baseline = week 0. 2nd MRI: week 8 after ERCP
  MRI baseline and follow-up will be assessed for dominant strictures to determine the reproducibility (capability to detect dominant strictures on both baseline and follow-up MRI) of dominant strictures that were not actively treated (dilated) with the invasive ERC. The assessment is performed by two independent radiologists, specialized in MRCP.

CONTACTS AND LOCATIONS:
Overall Officials: Cyriel Ponsioen, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Yes
After publication, the following documentation can be requested by qualified research groups:
  - Study protocol, statistical analysis plan and the clinical study report can be provided if a proper request is submitted.
  IPD will contain decoded and only essential data for the objective of this study. Data that will be available for sharing purposes will only include decoded demographic data. Furthermore, MRCP+ data that underlies the results in the publication will be available for sharing, e.g. MRCP+ metrics
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Until 5 years after publication
Access Criteria: Data sharing can be requested by qualified research groups. Requests will be evaluated by the following method:
  * The request is supposed to contain a clear objective and methodology. E.g., it must contain the objective to explore or validate the value of MRCP+ techniques. Furthermore, the study proposal could, for example, be a systematic review or meta-analysis.
  * The request will be reviewed by a dedicated research team of the MALD-study. This research team contains the PI, PhD student, involved gastro-enterologist and radiologist and representative of Perspectum Ltd.
  * If the request seems valid and the credibility of the requesting party is validated, data sharing agreement will be developed with the local research support team. To submit a request, contact t.e.middelburg@amsterdamumc.nl

REFERENCES:
- [Background] Ponsioen CY, Arnelo U, Bergquist A, Rauws EA, Paulsen V, Cantu P, Parzanese I, De Vries EM, van Munster KN, Said K, Chazouilleres O, Desaint B, Kemgang A, Farkkila M, Van der Merwe S, Van Steenbergen W, Marschall HU, Stotzer PO, Thorburn D, Pereira SP, Aabakken L. No Superiority of Stents vs Balloon Dilatation for Dominant Strictures in Patients With Primary Sclerosing Cholangitis. Gastroenterology. 2018 Sep;155(3):752-759.e5. doi: 10.1053/j.gastro.2018.05.034. Epub 2018 May 24. PMID 29803836
- [Background] Lazaridis KN, LaRusso NF. Primary Sclerosing Cholangitis. N Engl J Med. 2016 Sep 22;375(12):1161-70. doi: 10.1056/NEJMra1506330. No abstract available. PMID 27653566
- [Background] Zheng HH, Jiang XL. Increased risk of colorectal neoplasia in patients with primary sclerosing cholangitis and inflammatory bowel disease: a meta-analysis of 16 observational studies. Eur J Gastroenterol Hepatol. 2016 Apr;28(4):383-90. doi: 10.1097/MEG.0000000000000576. PMID 26938805
- [Background] Barner-Rasmussen N, Pukkala E, Jussila A, Farkkila M. Epidemiology, risk of malignancy and patient survival in primary sclerosing cholangitis: a population-based study in Finland. Scand J Gastroenterol. 2020 Jan;55(1):74-81. doi: 10.1080/00365521.2019.1707277. Epub 2020 Jan 4. PMID 31902255
- [Background] Boonstra K, Weersma RK, van Erpecum KJ, Rauws EA, Spanier BW, Poen AC, van Nieuwkerk KM, Drenth JP, Witteman BJ, Tuynman HA, Naber AH, Kingma PJ, van Buuren HR, van Hoek B, Vleggaar FP, van Geloven N, Beuers U, Ponsioen CY; EpiPSCPBC Study Group. Population-based epidemiology, malignancy risk, and outcome of primary sclerosing cholangitis. Hepatology. 2013 Dec;58(6):2045-55. doi: 10.1002/hep.26565. Epub 2013 Oct 17. PMID 23775876
- [Background] Hirschfield GM, Karlsen TH, Lindor KD, Adams DH. Primary sclerosing cholangitis. Lancet. 2013 Nov 9;382(9904):1587-99. doi: 10.1016/S0140-6736(13)60096-3. Epub 2013 Jun 28. PMID 23810223
- [Background] Ponsioen CY, Chapman RW, Chazouilleres O, Hirschfield GM, Karlsen TH, Lohse AW, Pinzani M, Schrumpf E, Trauner M, Gores GJ. Surrogate endpoints for clinical trials in primary sclerosing cholangitis: Review and results from an International PSC Study Group consensus process. Hepatology. 2016 Apr;63(4):1357-67. doi: 10.1002/hep.28256. Epub 2015 Dec 23. PMID 26418478
- [Background] Ponsioen CY, Reitsma JB, Boberg KM, Aabakken L, Rauws EA, Schrumpf E. Validation of a cholangiographic prognostic model in primary sclerosing cholangitis. Endoscopy. 2010 Sep;42(9):742-7. doi: 10.1055/s-0030-1255527. Epub 2010 Jul 9. PMID 20623444
- [Background] Lindor KD, Kowdley KV, Harrison ME; American College of Gastroenterology. ACG Clinical Guideline: Primary Sclerosing Cholangitis. Am J Gastroenterol. 2015 May;110(5):646-59; quiz 660. doi: 10.1038/ajg.2015.112. Epub 2015 Apr 14. PMID 25869391
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929
- [Background] Berstad AE, Aabakken L, Smith HJ, Aasen S, Boberg KM, Schrumpf E. Diagnostic accuracy of magnetic resonance and endoscopic retrograde cholangiography in primary sclerosing cholangitis. Clin Gastroenterol Hepatol. 2006 Apr;4(4):514-20. doi: 10.1016/j.cgh.2005.10.007. PMID 16616358
- [Background] Dave M, Elmunzer BJ, Dwamena BA, Higgins PD. Primary sclerosing cholangitis: meta-analysis of diagnostic performance of MR cholangiopancreatography. Radiology. 2010 Aug;256(2):387-96. doi: 10.1148/radiol.10091953. PMID 20656832
- [Background] Lunder AK, Hov JR, Borthne A, Gleditsch J, Johannesen G, Tveit K, Viktil E, Henriksen M, Hovde O, Huppertz-Hauss G, Hoie O, Hoivik ML, Monstad I, Solberg IC, Jahnsen J, Karlsen TH, Moum B, Vatn M, Negard A. Prevalence of Sclerosing Cholangitis Detected by Magnetic Resonance Cholangiography in Patients With Long-term Inflammatory Bowel Disease. Gastroenterology. 2016 Oct;151(4):660-669.e4. doi: 10.1053/j.gastro.2016.06.021. Epub 2016 Jun 21. PMID 27342213
- [Background] Zenouzi R, Welle CL, Venkatesh SK, Schramm C, Eaton JE. Magnetic Resonance Imaging in Primary Sclerosing Cholangitis-Current State and Future Directions. Semin Liver Dis. 2019 Jul;39(3):369-380. doi: 10.1055/s-0039-1687853. Epub 2019 Apr 30. PMID 31041791
- [Background] Goldfinger MH, Ridgway GR, Ferreira C, Langford CR, Cheng L, Kazimianec A, Borghetto A, Wright TG, Woodward G, Hassanali N, Nicholls RC, Simpson H, Waddell T, Vikal S, Mavar M, Rymell S, Wigley I, Jacobs J, Kelly M, Banerjee R, Brady JM. Quantitative MRCP Imaging: Accuracy, Repeatability, Reproducibility, and Cohort-Derived Normative Ranges. J Magn Reson Imaging. 2020 Sep;52(3):807-820. doi: 10.1002/jmri.27113. Epub 2020 Mar 8. PMID 32147892
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Tunnicliffe EM, Kelly C, Collier J, Wang LM, Fleming KA, Cobbold JF, Robson MD, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging for the assessment of non-alcoholic fatty liver disease severity. Liver Int. 2017 Jul;37(7):1065-1073. doi: 10.1111/liv.13284. Epub 2017 May 30. PMID 27778429
- [Background] Bradley CR, Cox EF, Scott RA, James MW, Kaye P, Aithal GP, Francis ST, Guha IN. Multi-organ assessment of compensated cirrhosis patients using quantitative magnetic resonance imaging. J Hepatol. 2018 Nov;69(5):1015-1024. doi: 10.1016/j.jhep.2018.05.037. Epub 2018 Jun 8. PMID 29886155
- [Background] Selvaraj EA, Culver EL, Coller J. Combination of quantitative MRCP and MRI demonstrates increased periductal iron-corrected T1 in primary sclerosing cholangitis. Gut. 2021;70:A155
- [Background] Ponsioen CY, Assis DN, Boberg KM, Bowlus CL, Deneau M, Thorburn D, Aabakken L, Farkkila M, Petersen B, Rupp C, Hubscher SG; PSC Study Group. Defining Primary Sclerosing Cholangitis: Results From an International Primary Sclerosing Cholangitis Study Group Consensus Process. Gastroenterology. 2021 Dec;161(6):1764-1775.e5. doi: 10.1053/j.gastro.2021.07.046. Epub 2021 Aug 10. No abstract available. PMID 34384749